CLINICAL TRIAL: NCT05787925
Title: The Efficacy of Adjunctive Oral Systemic Vitamin E Therapy on Salivary Nitric Oxide Level In Patients With Erosive Oral Lichen Planus (A Randomized Controlled Clinical Trial)
Brief Title: Adjunctive Oral Systemic Vitamin E Therapy on Salivary Nitric Oxide Level in Patients With Erosive Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0475-08
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Lichen Planus
MeSH Terms: conditions — Lichen Planus | interventions — Adrenal Cortex Hormones; Vitamin E

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical corticosteroid and Vitamin E (Experimental)
  Interventions: Drug: Topical corticosteroid and Vitamin E
- Topical corticosteroid (Active Comparator)
  Interventions: Drug: Topical corticosteroid

INTERVENTIONS:
Drug: Topical corticosteroid and Vitamin E — 26 patients who will administrate topical corticosteroid: triamcinolone acetonide 1% oral gel "Kenacort-A Orabase" * three times daily for 8 weeks applied after meals and at night with avoidance of foods and drinks for 30 minutes after the application. In addition to one capsule of 400 mg oral systemic vitamin E supplement* will be prescribed once daily at the morning
  Arms: Topical corticosteroid and Vitamin E
Drug: Topical corticosteroid — 26 patients will administrate topical corticosteroid: triamcinolone acetonide 1% oral gel "Kenacort-A Orabase" three times daily for 8 week that will be applied after meals and at night with avoidance of foods and drinks for 30 minutes after the application
  Arms: Topical corticosteroid

SUMMARY:
Oral lichen planus (OLP) is a chronic inflammatory disease affecting the skin, mucous membranes,s and rarely scalp and nails. It is a T-cell-mediated autoimmune disease. Traditional treatment for OLP is topical steroids commonly used to treat mild to moderately symptomatic lesions. Recent treatment modalities for oral lichen planus include micronutrients such as antioxidants including vitamin E that modify the immune system function. The aim of this study is to evaluate the efficacy of adjunctive oral systemic vitamin E therapy on salivary nitric oxide levels in patients with erosive oral lichen planus.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically and histopathologically confirmed of having erosive OLP according to modified WHO criteria.
* Patients with erosive OLP patients who will agree to take supplied medications.
* Ability to complete this trial.

Exclusion Criteria:

* OLP patients receiving any systemic treatment such as systemic steroids, other immunosuppressive drugs, or non-steroidal anti-inflammatory drugs on past 3 months.
* Pregnant and breast-feeding females.
* Patients suffering from systemic diseases.
* Patients with lesions showing any dysplastic changes in the biopsy specimen.
* Patients who are smoking and tobacco users in any form, will not be included.
* Patients with both lichenoid contact reaction and lichenoid drug reactions.
* Patients with cutaneous lichen planus lesions

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Change in oral lesion | At baseline,4th week and 8th week
  whole treatment response and the size of the oral lesions will be recorded using Thongprasom et al. scoring system, score 5 was assigned to patients having white striae with erosive areas >1 cm2, score 4 for patients with white striae and erosive areas <1 cm2, score 3 for those having white striae and atrophic areas >1 cm2, score 2 for those having white striae and atrophic areas <1 cm2, score 1 for those having only white striae, and score 0 for normal mucosa
Change in pain score | At baseline,4th week and 8th week
  At baseline, 4th week and 8th week after the treatment, burning sensation using Visual Analogue Scale (VAS) will be measured on a 10-point (0 = no symptoms, 10 = severe pain)

SECONDARY OUTCOMES:
Change in salivary nitric oxide | At baseline,4th week and 8th week
  Patients will be asked to rinse their mouth with 5 ml of normal saline for 3 min then tilt their head forward and expectorate saliva into a sterile beaker without swallowing. The saliva samples will be stored at -20 ºC till the time of analysis. It depends on the addition of Griess Reagents which convert nitrite into a deep purple azo compound; photometric measurement of the absorbance due to this azo chromophore accurately determines NO2-concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt